CLINICAL TRIAL: NCT05282082
Title: A Smart Surveillance Strategy for Carbapenem-resistant Pseudomonas Aeruginosa: the SAMPAN Study.
Brief Title: Carbapenem-resistant Pseudomonas Aeruginosa: the SAMPAN Study.
Acronym: SAMPAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, Medical coordinator Unit infection prevention, Erasmus Medical Center
Other Study IDs: 5025
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pseudomonas Aeruginosa; Colonization, Asymptomatic; Nosocomial Infection
MeSH Terms: conditions — Pseudomonas Infections; Asymptomatic Infections; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — CR-PA isolates will be collected and retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients at the moment of their admission to the hospital in one of the three cities: Swabs will be taken from patients who are willing to participate.
- Healthy volunteers living in "high-risk areas" in one of the three cities.: Swabs will be taken from healthy volunteers who are willing to participate.

SUMMARY:
Pseudomonas aeruginosa causes severe infections in hospitalized patients. The worldwide emergence of carbapenem-resistant P. aeruginosa (CR-PA) makes infections by these pathogens almost untreatable. The World Health Organization now ranks CR-PA highest in the list of 'urgent threats'. Information for action to prevent further emergence has to come from insight into sources and transmission routes through smart surveillance. At present, a smart surveillance strategy is not available for CR-PA. The aim of this project is to develop a globally-applicable smart surveillance strategy to guide action against the spread of CR-PA. Since P. aeruginosa prefers moist niches, we will focus on the human-water interface. First, highly-sensitive methods to detect CR-PA in specific environmental and human niches will be developed. Subsequently, CR-PA will be collected in three study sites with increasing prevalences of CR-PA, increasingly warmer climates, and different water situations: Rotterdam (The Netherlands), Rome (Italy), Jakarta (Indonesia). CR-PA will be searched for in a variety of niches in the environment outside and inside the hospital, and in healthy humans and hospitalized patients. Whole genome sequencing will be performed to compare the CR-PA from different sources and identify transmission routes. Our project will provide insight into the relative contribution of the different potential reservoirs of CR-PA to its spread in different settings which will be used for the development of a globally-applicable surveillance strategy for CR-PA to guide preventive actions.

ELIGIBILITY:
Inclusion Criteria healthy individuals:

* All healthy individuals living in a "high-risk area" in Rotterdam, Rome or Jakarta.

Exclusion Criteria healthy individuals:

* No signed consent sheet

Inclusion Criteria patients:

* Must be aged 18 years or older;
* Should be capable of providing answers to the questions in the questionnaire by himself/herself;
* Should have a minimum expected length of stay of at least 24 hours;
* Inclusion only once during the sampling year.

Exclusion Criteria patients:

* Cystic fibrosis patients
* No signed consent sheet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers are individuals living in "high-risk areas" in one of the three cities. "High-risk areas" are areas that we expect to have a high prevalence of CR-PA which may affect humans.
  Patients will be included at the moment of their admission to the hospital in one of the three cities. The three participating hospitals are all university hospitals.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalences of CR-PA in samples taken from healthy persons and patients at the moment of their admission to the hospital in the three cities. | 2023/2024

SECONDARY OUTCOMES:
Risk factors for carriage of CR-PA in healthy persons and patients. | 2023/2024

CONTACTS AND LOCATIONS:
Locations (3):
- Dr Cipto Mangunkusumo General Hospital, Jakarta, Indonesia
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes